CLINICAL TRIAL: NCT03204890
Title: Transcutaneous Posterior Tibial Nerve Stimulation (TPTNS) for Treating Patients With Premature Ejaculation. Phase II Clinical Trial
Brief Title: TPTNS for Treating Patients With Premature Ejaculation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Medical Group (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BMGC-2
Record Dates: First submitted 2017-06-28; First posted 2017-07-02 (Actual); Results first posted 2024-04-15 (Actual); Last update posted 2024-04-15 (Actual); Status verified 2023-10

CONDITIONS: Premature Ejaculation
MeSH Terms: conditions — Premature Ejaculation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TPTNS (Experimental): Transcutaneous Posterior Tibial Nerve Stimulation
  Interventions: Other: Transcutaneous Posterior Tibial Nerve Stimulation

INTERVENTIONS:
Other: Transcutaneous Posterior Tibial Nerve Stimulation — Three (3) sessions per week for twelve (12) consecutive weeks, with a duration of 30 minutes each, with the application of 20 Hertz with a pulse amplitude of 200 MI sec. in each session. The intensity will be applied individually for each patient depending on the tolerance of the individual. In each session, it is normal to have plantar flexion of the foot and flexion of the first toe, and after the session and particularly during the first sessions there is the possibility of muscle pain, which should be tolerable.

SUMMARY:
Background: Transcutaneous posterior tibial nerve stimulation is an effective therapy for controlling urinary incontinence. Premature ejaculation (PE) and urinary incontinence are anatomically and physio-pathologically similar. Based on this, the use of this therapy is considered to be viable for the control of PE.

Objective: To evaluate the efficacy of transcutaneous posterior tibial nerve electrostimulation for the ejaculatory reflex.

Patients and Methods: Phase II clinical trial. Patients with a diagnosis of premature ejaculation who are treated at the Colombia Boston Medical Group clinic will be included. The participants will receive 3 transcutaneous posterior tibial nerve stimulation therapies per week for 12 weeks. The IELT (Intravaginal ejaculatory latency time) and the PEDT (Premature Ejaculatory Diagnosis Tool) scale will be evaluated on week 6, at the end of treatment, and three months after completing the protocol.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age and less than 50 years of age with no cardiovascular risk factor other than age.
* Having been diagnosed with primary premature ejaculation according to the American Psychiatric Society's Diagnostic and Statistical Manual.
* Agreeing to participate and providing signed informed consent.
* Stable relationship for over 6 months, with frequent intercourse at least once per week.

Exclusion Criteria:

* Diagnosis of erectile dysfunction according to the International Index Function Erectile (IIFE-5) (score under 21).
* A premature ejaculatory diagnosis tool (PEDT) score under 8.
* Use of treatment for premature ejaculation during the study or over the 6 months prior to beginning the study.
* Use of pacemaker or heart defibrillator.
* Epilepsy or convulsions
* Venous insufficiency (varices) or cutaneous wounds or injuries on the lower extremities.
* Congenital or acquired anatomical abnormalities of the penis.
* Taking medications that affect ejaculation control, including psychiatric medications, opioid analgesics, and medications for pathologies of the prostate such as alpha-blockers.
* Psychological or psychiatric disorders that prevent the patient from undergoing the treatment or recording the measurements as established.
* Difficulty going to the clinic 3 times per week as required by the protocol.
* Patients with pre-coital premature ejaculation.
* Use of barrier contraceptive methods or local anesthetics.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2017-06-14 (Actual); Primary Completion 2018-01-15 (Actual); Study Completion 2018-10-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: José P Saffon, Doctor, Principal Investigator — Boston Medical Group
Locations (1):
- Boston Medical Group Colombia, Bogotá, Cundinamarca, Colombia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Ninety subjects with premature ejaculation were invited to participate in the study. Twenty-six men fulfilled the selection criteria and were enrolled between June 14, 2017 and March 14, 2018, in a specialized institute.
Pre-assignment Details: Fourteen participants had an IELT value >1 min during the evaluation with a stopwatch in the 2 weeks prior to the start of therapy and were excluded from the study.
Period: Overall Study
Arm/Group | TPTNS
Started | 12
Completed | 11
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | TPTNS
Number analyzed (Participants) | 12
Age, Customized [Median (Full Range); unit: years] | 30 [21 to 49]
Sex/Gender, Customized [Number; unit: participants]
  Men | 12
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Colombia | 12
Baseline Intravaginal ejaculation latency time (IELT) [Median (Full Range); unit: seconds] — Time in seconds between the start of vaginal intromission and the start of intravaginal ejaculation
  seconds | 30 [3 to 180]
Premature Ejaculation Diagnostic Tool (PEDT) score [Median (Full Range); unit: units on a scale] — The premature ejaculation diagnostic tool (PEDT), is a questionnaire for the diagnosis of premature ejaculation. The questionnaire has 5 questions and each of them scores from 0 to 4. The score is the sum of all the answers (range 0-20), with higher scores suggesting more difficulties with premature ejaculation. A score ≥11 points suggested the presence of premature ejaculation.
  units on a scale | 16 [11 to 20]

OUTCOME MEASURES:

1. Primary Outcome: Clinical Improvement
Description: Number of patients with clinical improvement of premature ejaculation, defined as a tripling of the baseline time (without treatment), as measured by the IELT (intravaginal ejaculation latency time)
Time Frame: Three months after completion.
Measure: Count of Participants; unit: Participants
Arm/Group | TPTNS
Number analyzed (Participants) | 11
Participants | 8

2. Secondary Outcome: Change in the Basal PDET Score
Description: The premature ejaculation diagnostic tool (PEDT), is a questionnaire for the diagnosis of premature ejaculation. The questionnaire has 5 questions and each of them scores from 0 to 4. The score is the sum of all the answers (range 0-20), with higher scores suggesting more difficulties with premature ejaculation. A score ≥11 points suggested the presence of premature ejaculation. This outcome indicates the number of patients who decrease their initial PEDT score after 3 months after completing treatment.
Time Frame: Three months after completion.
Measure: Number; unit: participants
Arm/Group | TPTNS
Number analyzed (Participants) | 11
participants | 7

3. Secondary Outcome: Magnitude of the Change in the PEDT Score
Description: The premature ejaculation diagnostic tool (PEDT), is a questionnaire for the diagnosis of premature ejaculation. The questionnaire has 5 questions and each of them scores from 0 to 4. The score is the sum of all the answers (range 0-20), with higher scores suggesting more difficulties with premature ejaculation. A score ≥11 points suggested the presence of premature ejaculation. This outcome indicates the average change that patients had in their PEDT score at baseline, 3 months after completing treatment.
Time Frame: Three months after completion.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | TPTNS
Number analyzed (Participants) | 12
score on a scale | 10.5 (5.2)

4. Secondary Outcome: Frequency of Adverse Events
Description: Number of patients with adverse events or side effects with the therapy
Time Frame: up to 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | TPTNS
Number analyzed (Participants) | 11
Participants | 2

ADVERSE EVENTS:
Time Frame: 9 months
Arm/Group | TPTNS
All-Cause Mortality (participants affected / at risk) | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11
Other Adverse Events (participants affected / at risk) | 2/11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TPTNS (N=11)
Not serious (Gastrointestinal disorders) | 1 (1) — Constipation
Not seriuos (Skin and subcutaneous tissue disorders) | 1 (1) — warmth sensation in leg

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2017-06-30): https://cdn.clinicaltrials.gov/large-docs/90/NCT03204890/Prot_SAP_ICF_000.pdf